CLINICAL TRIAL: NCT05802680
Title: Neurocognitive Effects of Non-Invasive Near-Infrared Light Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Francisco Gonzalez-Lima, PhD, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019080005
Record Dates: First submitted 2023-03-20; First posted 2023-04-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention Difficulties; Attention Deficit; Cognitive Deficit; Wellness
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sham-tPBM, non-ADHD (Sham Comparator): Participants with no medical diagnosis of ADHD will be exposed to the same conditions as treated participants, with the exception that the infrared light will be turned off (sham condition).
  Interventions: Device: Sham transcranial photobiomodulation
- Sham-tPBM, ADHD (Sham Comparator): Participants with a medical diagnosis of ADHD will be exposed to the same conditions as treated participants, with the exception that the infrared light will be turned off (sham condition).
  Interventions: Device: Sham transcranial photobiomodulation
- tPBM, non-ADHD (Experimental): Participants with no medical diagnosis of ADHD will be exposed to the same conditions as sham participants, with the exception that the infrared light will be turned on (treated condition).
  Interventions: Device: Transcranial photobiomodulation
- tPBM, ADHD (Experimental): Participants with a medical diagnosis of ADHD will be exposed to the same conditions as sham participants, with the exception that the infrared light will be turned on (treated condition).
  Interventions: Device: Transcranial photobiomodulation

INTERVENTIONS:
Device: Transcranial photobiomodulation — Administration of Sham or 1064 (+/- 50) nanometers tPBM
  Arms: tPBM, ADHD; tPBM, non-ADHD
Device: Sham transcranial photobiomodulation — Sham treatment
  Arms: Sham-tPBM, ADHD; Sham-tPBM, non-ADHD

SUMMARY:
Inattentiveness and impulsivity in healthy adults and individuals with attention deficit hyperactivity disorder (ADHD) diminish these individuals' quality of life. Cortical hypometabolism has been hypothesized to contribute to inattentiveness in ADHD. Transcranial photobiomodulation (tPBM) is a safe and non-invasive modality for activation of the prefrontal cortex. tPBM in healthy adults has been shown to augment brain oxygenation, cognition, and mood. The cognition-enhancing effect of tPBM on sustained attention in adults with ADHD remains unstudied. The investigators will evaluate whether tPBM administration to adults with and without ADHD can improve their attention. Each participant will be screened for eighteen criteria based on the Diagnostic and Statistical Manual (DSM-IV, text revised), using the validated instrument Adult ADHD Self-Report Scale (ASRS-v1.1). Blinded participants will be randomized into (I) Active-tPBM or (II) Sham-tPBM groups. After undergoing an 8-minute administration of Sham or 1064 nm tPBM to the lateral and medial right prefrontal cortex, each participant will complete a 14-minute, computer-based Conner's continuous performance task-3 (CPT-3). The investigators will examine whether adults with and without ADHD who receive Active-tPBM improve in measures of inattention, impulsivity, sustained attention, or vigilance compared to the Sham-tPBM group. Cognitive assessments of attention like the CPT-3 may evaluate the efficacy of tPBM to increase cortical metabolism in healthy adults and individuals with conditions like ADHD. The investigators anticipate their investigation will be a starting point for more sophisticated studies that focus on the implications of tPBM on cognition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Continuous Performance Task | Up to two months
  Measure of inattention, impulsivity, sustained attention, vigilance

SECONDARY OUTCOMES:
Functional near-infrared spectroscopy | Up to two months
  Resting state and activational state using a memory task

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Barrett, Ph.D., Study Director — University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared? Individual participant data that underlie the results reported in this study, after deidentification (text, tables, figures, and appendices).
  A data dictionary, including a description of the variables and types of data, collected for each individual, will be provided. This data will include anonymized individual participant demographic information and all outcome variables (continuous performance task, spectroscopy data).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: The raw data will be made available by the researchers upon reasonable request by any qualified doctoral researcher (PhD, MD). They will be granted access by contacting the corresponding author/principal investigator (F. Gonzalez-Lima, gonzalezlima@utexas.edu).
  It will be made available to qualified researchers whose proposed use of the data has been approved by an independent review committee (Institutional Review Board) identified for the purpose of individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months, the data will be available in our University's shared network drive, but without investigator support other than deposited metadata.
URL: https://labs.la.utexas.edu/gonzalez-lima/